CLINICAL TRIAL: NCT05396053
Title: Mirror Therapy Versus CIMT Improves Hand Strength and Function in Children With Unilateral Cerebral Palsy
Brief Title: Mirror Therapy Versus CIMT on Hand Function in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Mohamed A. Abdel Ghafar, Associate Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mirror Therapy
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Hemiplegic Cerebral Palsy; Mirror Hands
Keywords: Mirror therapy; Hand function; Grip strength
MeSH Terms: interventions — Exercise Therapy; Mirror Movement Therapy; Constraint Induced Movement Therapy

STUDY DESIGN:
Intervention Model Description: Study (2 groups) and control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): A traditional physical therapy program
  Interventions: Other: Physical therapy exercises
- Study 1 (Experimental): Mirror therapy plus traditional physical therapy program
  Interventions: Other: Physical therapy exercises; Other: Mirror therapy
- Study 2 (Experimental): Constraint-induced movement therapy plus traditional
  Interventions: Other: Physical therapy exercises; Other: Constraint Induced Movement Therapy

INTERVENTIONS:
Other: Physical therapy exercises — Three times a week for 12 weeks.
Other: Mirror therapy — Three times a week for 12 weeks.
  Arms: Study 1
Other: Constraint Induced Movement Therapy — Three times a week for 12 weeks.
  Arms: Study 2

SUMMARY:
The aim is to investigate the effect of mirror therapy on hand functions in children with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Hemiplegic cerebral palsy (HCP) is a form of paralysis that affects motor performance and muscle tone on one side of the body. Spastic hemiplegia CP is the second form of cerebral palsy in premature infants, affecting one side of the body's limbs. Hand and upper limb dysfunction cause problems in half of the children with cerebral palsy. Mirror therapy is a growingly recognized new treatment option for hemiplegic cerebral palsy. While upper extremity involvement in hemiplegic CP and the residual effects are more severe, there is limited evidence of the efficacy of mirror treatment in children with hemiplegic CP

ELIGIBILITY:
Inclusion Criteria:

* Spasticity grade 1 or 1+ based on the modified Ashworth scale
* Able to understand and follow instructions

Exclusion Criteria:

* Cognitive impairment
* Orthopedic dysfunction
* Impairment in visual acuity
* Children who are unable to pay attention during the treatment period

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 12 weeks
  Change of hand strength by using Hand Dynamometer
Hand function | 12 weeks
  Change of hand function skills by using Box and block test
Fine Motor skills | 12 weeks
  Change of fine motor skills score by using Peabody

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Abdel Ghafar, Ph.D, Principal Investigator — Batterjee Medical College
Locations (2):
- Saudi Arabia (2):
  - Batterjee Medical College, Jeddah
  - Local physical rehabilitation centers, Jeddah